CLINICAL TRIAL: NCT01654575
Title: Randomized Controlled Trial Using Methotrexate for Knee Osteoarthritis
Brief Title: Methotrexate in Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, Professor of Rheumatology, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: alexmed116662981
Record Dates: First submitted 2012-07-26; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Osteoarthritis
Keywords: Methotrexate; Knee Osteoarthritis; Synovitis; Pain reduction; Function scores
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Synovitis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Experimental): 25mg/week orally
  Interventions: Drug: Methotrexate
- Placebo (Active Comparator): Placebo-"sugar tablets" identical in colour and shape to methotrexate given once a week for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 25mg/week for 16 weeks
  Arms: Methotrexate
Drug: Placebo — Placebo tablets once a week for 16 weeks
  Arms: Placebo

SUMMARY:
Osteoarthritis (OA) is a common disabling condition, for which no effective therapy currently exists.Synovitis is commonly demonstrated in knee OA imaging. Methotrexate (MTX) helps to decrease synovitis in many inflammatory joint diseases, particularly rheumatoid arthritis.Accordingly,the aim of the present study was to assess the efficacy of MTX in decreasing pain and inflammation.Eighty-eight patients with clinical and radiographic criteria of primary knee OA with knee pain, were included in this study.Patients meeting the eligibility criteria were randomized in a 1:1 ratio to receive either 25mg/week oral MTX(n=44)or placebo(n=44)for 16 weeks. The primary outcome measure was pain reduction and secondary outcome measures included improvements in physical function scores.There was a statistically significant reduction in pain and improvement in function in the MTX group compared to the placebo group at 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis
* pain not responding to the usual therapy
* synovitis

Exclusion Criteria:

* any other inflammatory conditions,
* hepatic and renal insufficiency

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 4 months
Pain reduction | 16 weeks

SECONDARY OUTCOMES:
Improvement in physical function scores | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abou-Raya, MD, Study Director — University of Alexandria
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt